CLINICAL TRIAL: NCT02719522
Title: Pipeline Flex With SHield Technology Embolization - An International MulticEnter ObservationaL Post Market StuDy of Treated Intra Cranial Aneurysms (SHIELD)
Brief Title: Pipeline Flex With SHield Technology Embolization - An International MulticEnter ObservationaL Post Market StuDy
Acronym: SHIELD
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-PED-10
Record Dates: First submitted 2016-02-24; First posted 2016-03-25 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: Pipeline™ Flex Embolization Device with Shield Technology™ — Pipeline™ Flex Embolization Device with Shield Technology™ utilizes a phosphorylcholine (PC) surface treatment to the implant combined with the PFED delivery system. The Shield Technology™ surface treatment applied to the implant is an inert polymer material created to mimic the outer membrane of a human red blood cell.
  The Pipeline™ Flex Embolization Device with Shield Technology™ is intended for endovascular embolization of cerebral aneurysms and is designed to be placed across the opening (or 'neck') of a brain aneurysm and redirect blood flow away from the aneurysm, causing the blood within the aneurysm to clot.

SUMMARY:
This is a prospective, single-arm, multi-center post-market observational study assessing the performance of the Pipeline™ Flex Embolization Device with Shield Technology™ in subjects undergoing treatment for intracranial aneurysms in a large real-world, post-market setting.

DETAILED DESCRIPTION:
Eligible subjects will be treated with the Pipeline™ Flex Embolization Device with Shield Technology™.

Subjects will undergo standard of care follow-up visits. Data generated per standard of care will be collected for 1 year beyond the index procedure.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402 (j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402 (j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written Data Release Form (DRF) or informed consent using the Institutional Review Board (IRB)/ Ethic Committee (EC)-approved consent form and agrees to comply with protocol requirements.
* At least 18 years of age.
* Subject has already been selected for flow diversion therapy as the appropriate treatment.
* Subject has a target IA that has a parent vessel with diameter 1.5-5.0 mm distal/proximal to the target IA.

Exclusion Criteria:

* Major surgery including endovascular procedures within the past 30 days.
* Subject with target IA located in the basilar artery
* Subject with anatomy not appropriate for endovascular treatment due to severe intracranial vessel tortuosity or stenosis determined from baseline or pre-procedure imaging, or a history of intracranial vasospasm not responsive to medical therapy.
* Stent is in place in the parent artery at the target IA location.
* Subject with an acutely (within 30 days) ruptured aneurysm with a Hunt and Hess grade of 4 or higher.
* Any known contraindication to treatment with the Pipeline™ Flex Embolization Device with Shield Technology™ per Instructions for Use.
* The investigator determines that the health of the subject or the validity of the study outcomes (e.g., high risk of neurologic events, conditions that may increase the chance of stroke, worsening of clinical condition in the last 30 days) may be compromised by the subject's enrollment.
* Pregnant or breast-feeding women or women who wish to become pregnant during the length of study participation.
* Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from Medtronic.
* Legal incapacity or evidence that a subject cannot understand the purpose and risks of the study or inability to comply fully with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have an intracranial aneurysm (IA). The Pipeline™ Flex Embolization Device with Shield Technology™ will be used according to its Instructions for Use and its intended use during the treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Lamin, Study Chair — The Queen Elizabeth Hospital
Locations (21):
- Gold Coast University Hospital, Southport, Australia
- Rigshospitalet, Copenhagen, Denmark
- Turun Yliopistollinen keskussairaala, Turku, Finland
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Centrum, Berlin
  - Alfried Krupp Krankenhaus, Essen
  - Universitätsklinikums Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
- Hellenic Airforce Hospital, Athens, Greece
- Országos Klinikai Idegtudományi Intézet, Budapest, Hungary
- Hadassah Medical Organization, Jerusalem, Israel
- Italy (2):
  - Ospedale M. Bufalini, Cesena
  - Istituto Neurologico Carlo Besta, Milan
- Spain (5):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available

REFERENCES:
- [Background] Nelson PK, Lylyk P, Szikora I, Wetzel SG, Wanke I, Fiorella D. The pipeline embolization device for the intracranial treatment of aneurysms trial. AJNR Am J Neuroradiol. 2011 Jan;32(1):34-40. doi: 10.3174/ajnr.A2421. Epub 2010 Dec 9. PMID 21148256
- [Background] Becske T, Kallmes DF, Saatci I, McDougall CG, Szikora I, Lanzino G, Moran CJ, Woo HH, Lopes DK, Berez AL, Cher DJ, Siddiqui AH, Levy EI, Albuquerque FC, Fiorella DJ, Berentei Z, Marosfoi M, Cekirge SH, Nelson PK. Pipeline for uncoilable or failed aneurysms: results from a multicenter clinical trial. Radiology. 2013 Jun;267(3):858-68. doi: 10.1148/radiol.13120099. Epub 2013 Feb 15. PMID 23418004
- [Background] Kallmes DF, Hanel R, Lopes D, Boccardi E, Bonafe A, Cekirge S, Fiorella D, Jabbour P, Levy E, McDougall C, Siddiqui A, Szikora I, Woo H, Albuquerque F, Bozorgchami H, Dashti SR, Delgado Almandoz JE, Kelly ME, Turner R 4th, Woodward BK, Brinjikji W, Lanzino G, Lylyk P. International retrospective study of the pipeline embolization device: a multicenter aneurysm treatment study. AJNR Am J Neuroradiol. 2015 Jan;36(1):108-15. doi: 10.3174/ajnr.A4111. Epub 2014 Oct 29. PMID 25355814
- [Background] Chitale R, Gonzalez LF, Randazzo C, Dumont AS, Tjoumakaris S, Rosenwasser R, Chalouhi N, Gordon D, Jabbour P. Single center experience with pipeline stent: feasibility, technique, and complications. Neurosurgery. 2012 Sep;71(3):679-91; discussion 691. doi: 10.1227/NEU.0b013e318260fe86. PMID 22653389
- [Background] Saatci I, Yavuz K, Ozer C, Geyik S, Cekirge HS. Treatment of intracranial aneurysms using the pipeline flow-diverter embolization device: a single-center experience with long-term follow-up results. AJNR Am J Neuroradiol. 2012 Sep;33(8):1436-46. doi: 10.3174/ajnr.A3246. Epub 2012 Jul 19. PMID 22821921
- [Background] Kan P, Siddiqui AH, Veznedaroglu E, Liebman KM, Binning MJ, Dumont TM, Ogilvy CS, Gaughen JR Jr, Mocco J, Velat GJ, Ringer AJ, Welch BG, Horowitz MB, Snyder KV, Hopkins LN, Levy EI. Early postmarket results after treatment of intracranial aneurysms with the pipeline embolization device: a U.S. multicenter experience. Neurosurgery. 2012 Dec;71(6):1080-7; discussion 1087-8. doi: 10.1227/NEU.0b013e31827060d9. PMID 22948199
- [Background] Yu SC, Kwok CK, Cheng PW, Chan KY, Lau SS, Lui WM, Leung KM, Lee R, Cheng HK, Cheung YL, Chan CM, Wong GK, Hui JW, Wong YC, Tan CB, Poon WL, Pang KY, Wong AK, Fung KH. Intracranial aneurysms: midterm outcome of pipeline embolization device--a prospective study in 143 patients with 178 aneurysms. Radiology. 2012 Dec;265(3):893-901. doi: 10.1148/radiol.12120422. Epub 2012 Sep 20. PMID 22996749
- [Background] McAuliffe W, Wycoco V, Rice H, Phatouros C, Singh TJ, Wenderoth J. Immediate and midterm results following treatment of unruptured intracranial aneurysms with the pipeline embolization device. AJNR Am J Neuroradiol. 2012 Jan;33(1):164-70. doi: 10.3174/ajnr.A2727. Epub 2011 Oct 6. PMID 21979492
- [Background] Skukalek SL, Winkler AM, Kang J, Dion JE, Cawley CM, Webb A, Dannenbaum MJ, Schuette AJ, Asbury B, Tong FC. Effect of antiplatelet therapy and platelet function testing on hemorrhagic and thrombotic complications in patients with cerebral aneurysms treated with the pipeline embolization device: a review and meta-analysis. J Neurointerv Surg. 2016 Jan;8(1):58-65. doi: 10.1136/neurintsurg-2014-011145. Epub 2014 Nov 10. PMID 25385746
- [Derived] Rice H, Martinez Galdamez M, Holtmannspotter M, Spelle L, Lagios K, Ruggiero M, Vega P, Sonwalkar H, Chapot R, Lamin S. Periprocedural to 1-year safety and efficacy outcomes with the Pipeline Embolization Device with Shield technology for intracranial aneurysms: a prospective, post-market, multi-center study. J Neurointerv Surg. 2020 Nov;12(11):1107-1112. doi: 10.1136/neurintsurg-2020-015943. Epub 2020 Jun 1. PMID 32482834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients have been enrolled in 21 sites in EU, Australia and Israel between 24-Mar-2016 and 27-Sep-2017.
Groups:
- Intention to Treat (ITT): Includes all consented subjects in whom deployment of the Pipeline™ Shield device was attempted. For the ITT population, primary effectiveness endpoint analysis was based on Full Analysis Set (FAS) population and safety analysis was based on the ITT population.
Period: Overall Study
Arm/Group | Intention to Treat (ITT)
Started | 204 (In 1 consented subject, device deployment was not attempted due to significant arterial stenosis.)
Completed | 193
Not Completed | 11
Not completed — Implant Failure | 4
Not completed — Death | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.81)
Age, Customized [Count of Participants; unit: Participants]
  ≤60 years | 134
  > 60 years | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Greece | 21
  Hungary | 5
  Finland | 9
  Denmark | 3
  Italy | 26
  United Kingdom | 27
  Israel | 5
  Australia | 30
  France | 1
  Germany | 23
  Spain | 54

OUTCOME MEASURES:

1. Primary Outcome: Safety - Stroke/Death Occurrence
Description: Percentage (%) of Participants who experienced a major stroke in the territory supplied by the treated artery or neurological death post-procedure (1-year)
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients with event
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 204
percentage of patients with event | 3.23 [1.27 to 6.68]
Statistical Analysis 1: Comparison: Intention to Treat (ITT); The primary safety objective was to determine if the 2-sided 95% upper confidence interval of the primary safety endpoint was below the threshold of 15%. Missing safety data for subjects who were lost to FU without any evidence of a major stroke/death were imputed in the analysis using multiple imputation. Subjects who withdrew from the study prior to completion and had experienced a major stroke or death were counted towards the primary safety endpoint as having experienced the event; Test type: Superiority — The primary safety objective was to determine if the 2-sided 95% upper confidence interval of the primary safety endpoint was below the threshold of 15%; p < 0.001, Clopper-Pearson

2. Primary Outcome: Effectiveness - Aneurysm Occlusion
Description: Percentage (%) of Participants who have achieved complete aneurysm occlusion (defined as Raymond-Roy grade 1) without significant parent artery stenosis (≤ 50%) or retreatment of the target aneurysm post-procedure (1-year)
Time Frame: 1 year
Population: Primary effectiveness endpoint was analyzed specifically on subjects with successful device implantation (FAS population, N=200).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 200
percentage of patients | 71.67 [64.95 to 77.74]

3. Secondary Outcome: Safety - Stroke/Death Occurrence - 30 Days
Description: Percentage (%) of Participants who experienced a major stroke in the territory supplied by the treated artery or neurological death at 30 days post-procedure due to procedural complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 204
Participants | 6

4. Secondary Outcome: Safety - Intracerebral Hemorrhage (ICH)
Description: Percentage (%) of Participants who experienced a delayed intracerebral hemorrhage > 30 days post-procedure
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 204
Participants | 0

5. Secondary Outcome: Effectiveness - Deployment Rate
Description: Percentage (%) of Participants who have had a successful deployment of the device at the target site.
  A device is considered properly deployed when it covers the entire length of the aneurysm neck.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intention to Treat (ITT)
Number analyzed (Participants) | 204
Participants | 200

ADVERSE EVENTS:
Time Frame: Adverse Events have been collected through 1 year from study procedure.
Arm/Group | Intention to Treat (ITT)
All-Cause Mortality (participants affected / at risk) | 2/204
Serious Adverse Events (participants affected / at risk) | 44/204
Other Adverse Events (participants affected / at risk) | 74/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intention to Treat (ITT) (N=204)
Retinal artery occlusion (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2)
Cerebral microembolism (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Intracranial mass (Nervous system disorders) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3)
VIth nerve paralysis (Nervous system disorders) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 3 (3)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1)
Cranial nerve palsies multiple (Nervous system disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intention to Treat (ITT) (N=204)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 3 (3)
Visual impairment (Eye disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Vascular stent stenosis (General disorders) | 16 (16)
Contusion (Injury, poisoning and procedural complications) | 6 (6)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 6 (6)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 6 (6)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 4 (4)
Dysaesthesia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 11 (11)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3)
Polyneuropathy (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Vascular wall hypertrophy (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02719522/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT02719522/SAP_003.pdf